Ketamine and Propofol Combination Versus Propofol for Upper Gastrointestinal Endoscopy

Data Analysis Plan PI: Dr. Daniel Katz NCT02643979

Document Date: 12/20/2015

Ketamine and Propofol Combination Versus Propofol for Upper Gastrointestinal Endoscopy NCT02643979 12/20/2015

## Statistical Plan and Analysis:

All variables will be checked for normality via Shaprio Wilk Test. Our primary endpoint, since it is categorical in nature will be analyzed via chi square test. Each other categorical variable will be analyzed via chi square testing as well. For normally distributed variables, t-test will be used. For non-normally distributed variables non parametric tests such as Mann-Whitney-U and Wilcoxon Rank Sum will be used. Significance testing will all be two tailed, with a cutoff of 0.05 as the threshold for statistical significance.